CLINICAL TRIAL: NCT05775081
Title: Efficacy of Human Treated Dentine Matrix and Platelet Rich Fibrin in Induction of Root Formation of Non-Vital Immature Permanent Teeth
Brief Title: Treated Dentine Matrix and Platelet Rich Fibrin in Induction of Root Formation of Non-Vital Immature Permanent Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A07060721
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-09

CONDITIONS: Regenerative Endodontic Procedures; Necrotic Pulp
Keywords: Platelet rich fibrin, Treated dentine matrix
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated Dentine Matrix (TDM) (Experimental): Participants treated with TDM paste
  Interventions: Other: Regenerative endodontic procedues
- Platelet Rich Fibrin (PRF) (Experimental): Participants treated with PRF
  Interventions: Other: Regenerative endodontic procedues

INTERVENTIONS:
Other: Regenerative endodontic procedues — Treating non-vital immature permanent teeth with either treated dentine matrix paste or platelet rich fibrin

SUMMARY:
This study will be conducted to clinically evaluate the efficacy of human treated dentine matrix paste and Platelet rich fibrin (PRF) in induction of root formation of non-vital immature permanent teeth.

DETAILED DESCRIPTION:
A) Patient grouping:

Patients will be randomly allocated into 2 groups using sealed envelope method of randomization

Group (A):

Teeth to be treated by h-TDM paste (n=10).

Group (B):

Teeth to be treated by platelet rich fibrin (PRF) regeneration (n=10).

B) Procedures:

Diagnosis of pulp necrosis, clinical and radiographic examination. 11 For each patient, the protocol of treatment is composed of 7 sessions. The follow-up takes place over a 15 months' period. Day 0 is considered as the day of the first treatment session.

I- Day 0:

* Pre-operative Cone Beam Computed Tomography (CBCT) is taken at this visit.
* Calcium hydroxide canal conditioning for 2 weeks regardless of the treatment group. This is done in the following sequence:

  * Administration of local anesthesia, then rubber dam isolation.
  * Preparing an access cavity and establishing the working length by taking a radiograph with a file inserted into the root canal within 2 mm of the radiographic apex.
  * The canal is cleaned by irrigation with 1.25% sodium hypochlorite and the use of manual files. The cleaning and shaping are realized with files with a very light parietal action to avoid the canal widening and the weakening of the root walls. Above all, it consists in removing the pulp remnants.
  * Then, the canal is dried with paper point and can be filled with calcium hydroxide. Calcium hydroxide paste is prepared by mixing the calcium hydroxide powder and Barium Sulfate as a radio-opacifier mixed with sterile distilled water. A plug of calcium hydroxide is placed in the canal and condensed to the apical end of the root with a plugger. Other layers of calcium hydroxide are placed till complete canal filling.
  * The intracanal dressing quality is checked with a radiograph. The access cavity is temporarily sealed with a resin modified glass ionomer cement. This calcium hydroxide canal conditioning is performed for all patients to allow the complete disinfection.

II- Day 0+15:

This session starts with administration of local anesthesia, placement of a rubber dam and the removal of all the calcium hydroxide by copious saline irrigation. Then, treatment according to the assigned group:

Group A (h-TDM paste):

1. Preparation of h-TDM:

   Mentioned before.
2. Preparation of h-TDM paste:

Mentioned before. 3- Operative procedures:

* The h-TDM paste will be placed into the canal by sterile amalgam carrier and condensed to the apical end of the root with a plugger to create a 4 mm apical plug. Radiograph will be taken to verify proper placement of the mixture. Then, 1mm of MTA will be placed over this paste.
* Then, the access cavity will be filled with resin modified glass ionomer.

Group B (PRF regeneration):

13

* Ten ml of venous blood will be withdrawn from the child's forearm to a sterile test tube without anticoagulant and will be centrifuged in 3000 rpm for 10 minutes to prepare PRF, which appears as a membrane between the free plasma in the top and RBCs in the bottom of the tube.
* Platelet rich fibrin will be withdrawn from the test tube using sterile tweezer and put into sterile gauze and cut into small pieces using sterile scissor.
* Root canal will be copiously irrigated by sterile saline and dried with sterile paper points. Platelet rich fibrin small pieces will be condensed into the root canal till the apex using sterile plugger. Then, 2mm of MTA will be placed over the PRF till CEJ. Then, access cavity will be sealed by glass ionomer.

III- 3 months:

Clinical and radiographic control for all patients.

IV- 6 months:

Clinical and radiographic control for all patients.

V- 9 months:

Clinical and radiographic control for all patients.

VI- 12 months:

• Clinical and radiographic control for all patients.

VII- 15 months:

* Clinical and radiographic control for all patients.
* CBCT is taken at this visit. The x-rays of each patient are taken with the aid of film holder to be standardized and reproducible, so that they can be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 6-11 years presenting with a non-vital permanent immature tooth.

Exclusion Criteria:

* History of uncontrolled diabetes
* Immunosuppression
* Chronic systemic disease if a treatment is required
* Periodontal disease

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation | 15 months
  Clinically evaluating the efficacy of human treated dentine matrix paste and Platelet rich fibrin (PRF) in induction of root formation of non-vital immature permanent teeth.

SECONDARY OUTCOMES:
Radiographic evaluation | 15 months
  Radiographically evaluating the efficacy of human treated dentine matrix paste and Platelet rich fibrin (PRF) in induction of root formation of non-vital immature permanent teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Asal, MDS, Principal Investigator — Mansoura University; Ibrahim H Elkalla, PhD, Study Chair — Mansoura University; Yousry M Elhawary, PhD, Study Director — Mansoura University; Ashraf Y Alhsoainy, PhD, Study Director — Mansoura University
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No